CLINICAL TRIAL: NCT02582086
Title: A Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Safety and Efficacy of a Topical Natural Health Product for the Treatment of Herpes Labialis
Brief Title: Study of a New Topical Natural Health Product for the Treatment of Herpes Labialis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laboratoire Boreaderme Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15E-0601
Record Dates: First submitted 2015-10-16; First posted 2015-10-21 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Herpes Labialis
MeSH Terms: conditions — Herpes Labialis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BOR15001L7 Cream (Experimental): BOR15001L7 Cream with 5% 15019L0
  Interventions: Other: BOR15001L7
- Placebo Cream (Placebo Comparator): Placebo Cream
  Interventions: Other: Placebo

INTERVENTIONS:
Other: BOR15001L7 — Active cream with 5% 15019L0
  Arms: BOR15001L7 Cream
Other: Placebo — Placebo Cream with 0% 15019L0
  Arms: Placebo Cream

SUMMARY:
The aim of this study is to determine the safety and efficacy of a topical natural health product in comparison to placebo for the treatment of herpes labialis.

ELIGIBILITY:
Inclusion Criteria:

* Female and male, in good health, 18 years of age or older,
* With history of recurrent herpes labialis with at least twice a year during the past twenty-four months,
* Agreeing not to take another treatment against cold sore, nor anti-inflammatory, antibiotics and steroids,
* Cooperating in the study, able to be monitored at each visit, aware of the demands and duration of the controls, thus allowing perfect adherence to the established protocol,
* Must be willing and able to participate and to provide written informed consent,
* Female subjects of childbearing potential must have a negative pregnancy test at screening and agree to use a proper contraceptive method during the study.

Exclusion Criteria:

* Volunteers who refuse to introduce the product to be tested in its routine,
* With a history of hypersensitivity to the type of product to be tested (e.g., products that contain essential oil),
* Who have a history of eczema, topical dermatitis, psoriasis or significant skin anomalies on the areas to be tested,
* Who suffer from a serious illness or health problem or a critical or progressive disease,
* Who have taken prescription or over the counter medication that could affect skin characteristics or could bias the study (i.e. antibiotics, antihistamines, anti-inflammatories…) within 7 days prior to study beginning,
* Who have recently acquired or who currently have significant skin pigmentation, who frequent tanning salons or foresee exposure to the sun during the study,
* Who abuse alcohol, drugs and/or tobacco,
* Female subjects who are pregnant, breastfeeding or expecting to become pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Time to healing as assessed by the investigator | up to 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Evalulab Inc, Montreal, Quebec, Canada